CLINICAL TRIAL: NCT05717517
Title: Corneal Changes After Collagen Cross-linking ; Clinical and Oct Study
Brief Title: Collagen Cross-linking Clinical and Oct Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Aly, resident doctor, Assiut University
Other Study IDs: ant seg oct in cross linking
Record Dates: First submitted 2021-10-19; First posted 2023-02-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Corneal Ectasia of Both Eyes
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: anterior segment oct — ant segment oct before and after corneal collagen cross-linking
  Other Names: collagen cross linking

SUMMARY:
1. Assessment of corneal changes in AS-OCT after collagen cross-linking (corneal thickness and demarcation line).
2. Assessment of the effect of collagen cross-linking on best-corrected visual acuity

DETAILED DESCRIPTION:
Cross-linking of collagen refers to the ability of collagen fibrils to form strong chemical bonds with adjacent fibrils. In the cornea, collagen cross-linking occurs naturally with aging due to an oxidative deamination reaction that takes place within the end chains of the collagen. It has been hypothesized that this natural cross-linkage of collagen explains why keratectasia (corneal ectasia) often progresses most rapidly in adolescence or early adulthood but tends to stabilize in patients after middle-age.

Human studies of UV-induced corneal cross-linking began in 2003 in Dresden, and early results were promising. The initial pilot study enrolled 16 patients with rapidly progressing keratoconus and all of the patients stopped progressing after treatment. Additionally, 70% had flattening of their steep anterior corneal curvatures (decreases in average and maximum keratometric values), and 65% had an improvement in visual acuity. There were no reported complications.

Per the typical cross-linking protocol, 0.1% riboflavin solution with 20% dextran is added to the de-epithelialized cornea and then photoactivated with UV-A light at 365 nm with irradiance of 3 mW/cm2 for 30 minutes. The cornea is de-epithelialized to allow adequate penetration of riboflavin into the corneal stroma. Riboflavin acts as photosensitizer; it creates free radicals, forms new molecular crosslinks, and ultimately increases the cornea's mechanical strength.

Collagen cross-linking experienced a rapid transition from laboratory procedure to clinical intervention because of the method's apparent safety and broad array of potential applications. One such clinical application is the treatment of keratoconus which is a degenerative disorder of the eye associated with thinning and subsequent bulging of the cornea, causing poor vision. Collagen cross-linking stops the progression of keratoconus in patients with mild disease, presumably by strengthening the cornea and preventing further bulging.

Collagen cross-linking has also been used successfully in the treatment of pellucid marginal degeneration and to treat iatrogenic (postoperative) ectasia. Studies have shown that CXL causes a reduction in corneal edema and thickness with improvement in visual acuity in patients with bullous keratopathy due to different causes. However, these changes last for only about six months and due to this transient effect, CXL may only have a palliative role, if at all, for now.

The effect of cross linking can be assessed postoperatively clinically and also by some devices such as Ocular Response Analyzer (Reichert Inc., Buffalo, NY, USA). The depth of treatment can be measured by the demarcation line, which usually appears at 10 to 14 days after CXL and can be monitored using corneal topography and tomography.

Optical coherence tomography (OCT) is a modality that uses low-coherence interferometry to enable non-contact, in vivo imaging of ocular structures. Since its introduction, OCT imaging has become a key part of clinical evaluation of the cornea, and the anterior eye segment.

As improvements to the technology have increased, e.g. the speed and resolution of the images captured, the impact of anterior segment OCT (AS OCT) imaging on clinical practice, has been rapidly increasing and the clinical potential of the technique in evaluating the cornea had been realized. Specific to the cornea, AS OCT now allows us to image corneal layers and structures in greater detail i.e. epithelium, Bowman's layer, stroma, Descemet membrane and endothelium.

The AS OCT is extremely useful in studying anterior segment pathology through an edematous cornea such as in Descemet membrane detachments , corneal stroma itself and corneal infiltrates secondary to infections.

AS OCT is also useful in assessing changes in cornea postoperative including corneal changes after cross linking. The most widely reported change seen on cross-sectional OCT following CXL has been the appearance of a 'demarcation' line within the corneal stroma. This line has been postulated to represent the depth of the CXL treatment, separating the treated anterior stroma and untreated posterior stroma. The demarcation line is hyper-reflective when viewed with OCT, Scheimpflug imaging and on slit lamp biomicroscopy. OCT provides the ability to measure the depth of the demarcation line and has been used as an important outcome parameter when comparing various CXL protocols. The demarcation line usually fades by three months and, in some corneas, is replaced with faint, irregular, hyper-reflective lines in the deep stroma.

Other changes that can be noted on OCT images following CXL include increased reflectivity of the treated stroma, and the appearance of fainter, secondary stromal demarcation lines.

ELIGIBILITY:
Inclusion Criteria:

* patients with e corneal ectasia who are candidates for CXL.

Exclusion Criteria:

* patients with other corneal diseases not treated by collagen cross-linking
* corneal scarring.
* previous corneal surgeries (e.g intrastromal corneal ring segments)

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: patients who underwent classic corneal collagen cross-linking
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
corneal thickness after collagen cross linking OCT study | 12 months
  corneal thickness measurement in mm

SECONDARY OUTCOMES:
corneal demarcation line after collagen cross linking OCT study | 12 months
  measurement of the depth of demarcation line from tear film in mm

REFERENCES:
- [Background] Wollensak G, Spoerl E, Seiler T. Stress-strain measurements of human and porcine corneas after riboflavin-ultraviolet-A-induced cross-linking. J Cataract Refract Surg. 2003 Sep;29(9):1780-5. doi: 10.1016/s0886-3350(03)00407-3. PMID 14522301
- [Background] Raiskup F, Spoerl E. Corneal crosslinking with riboflavin and ultraviolet A. I. Principles. Ocul Surf. 2013 Apr;11(2):65-74. doi: 10.1016/j.jtos.2013.01.002. Epub 2013 Jan 24. PMID 23583042
- [Background] Brummer G, Littlechild S, McCall S, Zhang Y, Conrad GW. The role of nonenzymatic glycation and carbonyls in collagen cross-linking for the treatment of keratoconus. Invest Ophthalmol Vis Sci. 2011 Aug 11;52(9):6363-9. doi: 10.1167/iovs.11-7585. PMID 21724915
- [Background] Raiskup F, Terai N, Velika V, Sporl E. [Corneal Cross-Linking with Riboflavin and UVA in Keratoconus]. Klin Monbl Augenheilkd. 2016 Aug;233(8):938-44. doi: 10.1055/s-0042-102060. Epub 2016 Apr 7. German. PMID 27055493